CLINICAL TRIAL: NCT01569412
Title: Phase I/II, Open Label, Dose Escalating Study To Investigate Safety, Tolerability, And Preliminary Efficacy Of The Trifunctional Anti-HER-2/Neu x Anti-CD3 Antibody Ertumaxomab In Patients With HER-2/Neu Expressing (1+/SISH Positive, 2+ and 3+) Solid Tumors Progressing After Standard Therapy
Brief Title: Open Label, Dose Escalating Study With Ertumaxomab In Patients With HER-2/Neu Expressing Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Krankenhaus Nordwest (Other)
Responsible Party: Principal Investigator, Prof. Dr. S.E. Al-Batran, Principal Investigator, Krankenhaus Nordwest
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERTUSO
Record Dates: First submitted 2012-03-09; First posted 2012-04-03 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Her2/Neu Positive Advanced Solid Tumors
MeSH Terms: interventions — ertumaxomab

ARMS (1):
- Ertumaxomab (Experimental): Ertumaxomab administration during two treatment cycles will follow a predefined dose escalation scheme, consisting of 5 ascending doses per cycle with each infusion lasting 3 hours.
  Interventions: Biological: Ertumaxomab

INTERVENTIONS:
Biological: Ertumaxomab — trifunctional antibody, infusion i.v., increasing doses, up to 10 infusions

SUMMARY:
Patients with HER2/neu expressing solid tumors progressing after standard therapy will be treated with a so called trifunctional antibody (Ertumaxomab). The main objective of this trial is to find the maximum tolerated dose. Tolerability and Safety will be assessed as well as efficacy.

DETAILED DESCRIPTION:
This is an open label phase I/II study dose escalating study to investigate safety, tolerability, and preliminary efficacy of the trifunctional anti-HER2/neu x anti-CD3 antibody ertumaxomab in patients with HER2/neu (1+/SISH positive, 2+ and 3+) expressing solid tumors progressing after standard therapy. The primary objectives of the study is to assess the safety and tolerability of ertumaxomab in order to determine the maximum tolerated dose (MTD) and to establish a recommended dose (RD) for further development.

A maximum of ten infusions will be applicated.

Patients will be seen at baseline/screening, and then weekly for infusion and safety assessment with a break of 3 weeks after the 5th dose. Radiological tumor assessment will be performed every 6 weeks. Post-study follow-up will be completed every 8 weeks for up to one year.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form.
* Male or female patients aged ≥ 18 years and with a life expectancy of at least 4 months.
* Negative pregnancy test at screening (and not more than 72 hours prior to the first ertumaxomab infusion) for women of childbearing potential. Patients must agree to use adequate contraception during the study.
* Measurable disease, defined as at least one lesion that is measurable in one dimension.
* Solid HER2/neu positive tumors (1+/SISH positive, 2+, and 3+), histologically confirmed.
* Patients must have disease progression during or after standard therapy and/or are no longer feasible for approved therapies.
* Previous therapies must be discontinued at least 2 weeks (6 weeks in case mitomycin C) prior to administration of ertumaxomab and all treatment related toxicities must have resolved or decreased to common toxicity criteria (CTC) grade 1 (with the exception of alopecia and peripheral neuropathy).
* If patients have received HER2-targeting therapies, all HER2-targeting therapies must have been discontinued before study entry.
* Eastern Cooperative Oncology Group (ECOG) performance score of ≤ 2.
* Adequate hematological, liver and kidney function:
* Adequate recovery from prior systemic therapy.
* Patients capable to understand the purposes and risks of the study, and who are willing and able to participate in the study
* Left ventricular ejection fraction must be > 50% at echocardiography

Exclusion Criteria:

* Patients currently being treated with medication or anticonvulsants for brain or central nervous system metastases or patients that have documented radiologic evidence of active brain or central nervous system metastases within 12 weeks of study entry.
* Patients with a prior diagnosis of any other malignancy (unless cured by surgery or other appropriate treatments greater than 2 years before study entry). Patients with in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin may be included at any time.
* ≥ 5 preceding chemotherapies
* Documented acute or chronic infection or other concurrent non-malignant co morbidities that are uncontrolled, such as unstable or uncontrolled pectorial angina, myocardial infarction during the last 6 months, valvular heart disease that requires treatment, acute myocarditis or congestive heart failure (CHF, NYHA III or IV).
* Patients with a known human immunodeficiency virus, hepatitis B or hepatitis C positive status are excluded from participation in the study
* Any concurrent chemotherapy, radiotherapy (except for local radiation therapy for bone marrow metastasis), hormonal therapy, immunotherapy or corticoid therapy.
* Treatment with any investigational product within 2 weeks prior to first administration of ertumaxomab.
* Patients with documented autoimmune diseases.
* Known hypersensitivity to murine proteins and any other component of the drug.
* Abnormal organ or bone marrow function as defined below (any single parameter to fulfill condition):

  * ANC < 1.5 Gpt/l (1.5x109/L, 1500/mm3)
  * Hemoglobin <9.0 g/dl
  * Platelet count < 75Gpt/l (75x109/L, 75,000/mm³)
  * AST(SGOT)/ALT(SGPT) > 3 x upper limit of normal (ULN); or: in case of metastatic liver disease AST(SGOT)/ALT(SGPT) > 5 x ULN
  * Alkaline Phospatase > 2.5 x ULN
  * Serum (total) bilirubin > 1,5 x ULN for the institution; or in case of metastatic liver disease: Serum (total) bilirubin > 3 x ULN for the institution;
  * Serum creatinine > 1.5 x ULN
* Any other concurrent disease or medical conditions that are deemed to interfere with the conduct of the study as judged by the investigator.
* Known hypersensitivity to ertumaxomab and its analogues in general, or to any other component of the study drug formulation.
* Pregnant women, nursing mothers, lactating women, and women of child-bearing potential who are unwilling to use effective contraception (see above).
* Use of immune-suppressive agents for the past 4 weeks prior to the first administration of ertumaxomab. For regular use of systemic corticosteroids, patients should only be included after stepwise discontinuation to be free of steroids for a minimum of 7 days prior to first treatment.
* Unwilling or unable to follow protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose | every week until end of treatment (max. 108 days)

SECONDARY OUTCOMES:
Pharmacodynamic | weekly until end of treatment (max. 108 days)
  Determination of HAMA, Serum levels of cytokines IL2, 6, 8, TNF-alpha, IFN-gamma, Blood cell count (immune status), Humoral immune responses (autologous anti-EpCAM / anti-Her2neu antibodies), Identification of T memory cells
efficacy according to RECIST and immune related response criteria (irRC) | every 6 weeks until progression of disease
adverse events | weekly (max 108 days)
  incidence and intensity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, MD, Principal Investigator — Institute of Clinical Cancer Research (IKF), UCT - University Cancer Center, Frankfurt, Germany
Locations (1):
- Krankenhaus Nordwest, Frankfurt am Main, Germany

REFERENCES:
- [Derived] Haense N, Atmaca A, Pauligk C, Steinmetz K, Marme F, Haag GM, Rieger M, Ottmann OG, Ruf P, Lindhofer H, Al-Batran SE. A phase I trial of the trifunctional anti Her2 x anti CD3 antibody ertumaxomab in patients with advanced solid tumors. BMC Cancer. 2016 Jul 7;16:420. doi: 10.1186/s12885-016-2449-0. PMID 27387446